CLINICAL TRIAL: NCT04404426
Title: CACOLAC : Randomized Trial of Citrulline Administration in the Hospital Patient in Intensive Care for COVID-19 Acute Respiratory Distress Syndrome
Brief Title: CACOLAC : Citrulline Administration in the Hospital Patient in Intensive Care for COVID-19 Acute Respiratory Distress Syndrome
Acronym: CACOLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC20_9815_CACOLAC; CPP 1288 HPS1 (Other: CPP Ouest 6 (Brest)); 2020-A01189-30 (Other: ID RCB)
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: ARDS Secondary to COVID-19 Pneumonia
MeSH Terms: interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, placebo-controlled, randomized, double-blind, two-parallel study, specific enteral administration by citrulline in a subgroup of resuscitation patients admitted for ARDS secondary to COVID-19 pneumonia, at infectious risk nosocomial important because having biological stigmas of immunosuppression on admission and under invasive mechanical ventilation for a prolonged period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-citrulline (Experimental): Administration of citrulline enterally for 7 days
  Interventions: Dietary Supplement: L-citrulline
- Placebo (Placebo Comparator): Administration of placeboenterally for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — Administration of citrulline enterally for 7 days.
  Arms: L-citrulline
Other: Placebo — Administration of placebo (water) enterally for 7 days
  Arms: Placebo

SUMMARY:
Respiratory involvement of SARS-CoV2 leads to acute respiratory distress syndrome (ARDS) and significant immunosuppression (lymphopenia) exposing patients to long ventilation duration and late mortality linked to the acquisition of nosocomial infections.

Lymphopenia characteristic of severe forms of ARDS secondary to SARS-CoV2 infection may be linked to expansion of MDSCs and arginine depletion of lymphocytes.

Severe forms of COVID-19 pneumonitis are marked by persistent ARDS with acquisition of nosocomial infections as well as by prolonged lymphocytic dysfunction associated with the emergence of MDSC.

It has been found in intensive care patients hypoargininaemia, associated with the persistence of organ dysfunction (evaluated by the SOFA score), the occurrence of nosocomial infections and mortality. Also, it has been demonstrated that in these patients, the enteral administration of ARG was not deleterious and increased the synthesis of ornithine, suggesting a preferential use of ARG by the arginase route, without significant increase in argininaemia nor effect on immune functions. L-citrulline (CIT), an endogenous precursor of ARG, is an interesting alternative to increase the availability of ARG. Recent data demonstrate that the administration of CIT in intensive care is not deleterious and that it very significantly reduces mortality in an animal model of sepsis, corrects hypoargininemia, with convincing data on immunological parameters such as lymphopenia, which is associated with mortality, organ dysfunction and the occurrence of nosocomial infections. The availability of ARG directly impacts the mitochondrial metabolism of T lymphocytes and their function. The hypothesis is therefore that CIT supplementation is more effective than the administration of ARG to correct hypoargininaemia, decrease lymphocyte dysfunction, correct immunosuppression and organ dysfunction in septic patients admitted to intensive care.

The main objective is to show that, in patients hospitalized in intensive care for ARDS secondary to COVID-19 pneumonia, the group of patients receiving L-citrulline for 7 days, compared to the group receiving placebo, has a score of organ failure decreased on D7 (evaluated by the SOFA score) or by the last known SOFA score if the patient has died or been resuscitated.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Patients admitted for less than 48 hours in intensive care for ARDS under mechanical ventilation according to the Berlin criteria published in 2012 (JAMA);
* Origin of ARDS: COVID-19 pneumopathy confirmed by PCR (nasopharyngeal or tracheal sample);
* Life expectancy> 2 days;
* Affiliated to a social security scheme;
* Consent signed by the patient, the relative or the legal representative (except emergency procedure).

Exclusion Criteria:

* Pregnancy or breastfeeding in progress;
* State of immunosuppression defined by at least one of these criteria: continuous administration of steroids at any dose for more than a month before hospitalization, steroids in high doses (> 15 mg / kg / day of methylprednisolone or equivalent), radiotherapy or chemotherapy in the previous year, proven humoral or cellular deficiency;
* Contraindication to enteral nutrition (2016 SRLF recommendations: "Enteral nutrition probably should not be used upstream of a high-flow digestive fistula in the event of intestinal obstruction, small ischemia or digestive hemorrhage active (Strong chord) ").
* Ongoing immunosuppressive therapy such as chemotherapy, cyclophosphamide, high dose corticosteroid therapy (> 15 mg / kg / day);
* Participation in intervention research on a drug, or intervention research that may impact the immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
SOFA | Day 8
  SOFA score for organ failures on D8 or last known SOFA score if the patient has died or been resuscitated

SECONDARY OUTCOMES:
Number and phenotype of lymphocytes | Days 1, 8 and 14
  Number and phenotype of lymphocytes on days 1, 8 and 14
HLA-DR | Days 1, 8 and 14
  Monocytic expression HLA-DR (Flow cytometry) on days 1, 8 and 14
Number of Myeloid-derived suppressor cells | Days 1, 8 and 14
  Number of Myeloid-derived suppressor cells (Flow cytometry) on days 1, 8 and 14
Plasma cytokines / chemokines | Days 1, 8 and 14
  Plasma cytokines / chemokines (IL-6, IL-8, IL-10, IL-7, CXCL10, G-CSF, TNF-alpha, IFN-β) at days 1, 8 and 14
Repertoire T | Days 1, 3, 8, 10 and 14
  Diversity of the repertoire T at days 1, 3, 8, 10 and 14
Lymphocyte T exhaustion | Days 1, 8 and 14
  T lymphocyte exhaustion: measurement of lymphocyte apoptosis and lymphocyte proliferation on days 1, 8 and 14
Mitochondrial activity | Days 1, 8 and 14
  Measurement of mitochondrial activity (measurement of the number of mitochondria and their membrane potential, measurement of the expression of Beclin1) on days 1, 8 and 14
Plasma amino acids | Days 1, 8 and 14
  Plasma amino acids (arginine and its metabolites (ornithine, glutamate, glutamine, citrulline, proline) and tryptophan / kynurenine) on days 1, 8 and 14
SOFA | Days 3, 7, 10 and 14
  SOFA score of organ failures on days 3, 7, 10 and 14
Duration of hospitalization in intensive care | Day 28
  Duration of hospitalization in intensive care (days), up to day 28 maximum
Duration of hospital stay in hospital | Day 28
  Duration of hospital stay in hospital (days), up to day 28 maximum
Duration of mechanical ventilation | Day 28
  Duration of mechanical ventilation (days), up to day 28 maximum
Mortality in intensive care on day 28 | Day 28
  Mortality in intensive care on day 28
Hospital mortality on day 28 | Day 28
  Hospital mortality on day 28
Measurement of the presence of SARS-CoV2 | Days 1, 8 and 14
  Measurement of the presence of SARS-CoV2 in the tracheal aspiration by PCR on days 1, 8 and 14
Nosocomial infections | D28
  Incidence of nosocomial infections during the intensive care unit (maximum D28). The diagnosis of nosocomial infections will be made according to the definitions of nosocomial infections of the CDC. An independent committee of experts will validate or not the infections
Number of days of exposure to each antibiotic per 1000 days of hospitalization | Day 28
  Number of days of exposure to each antibiotic per 1000 days of hospitalization (maximum day 28).

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Britanny, France

IPD SHARING:
Plan to Share IPD: Undecided